CLINICAL TRIAL: NCT01266291
Title: Sabril for Treatment of Adult Refractory Partial Seizures Symptomatic of Tuberous Sclerosis: An Open Label, Phase IV Prospective Safety and Tolerability Study
Brief Title: Sabril for Complex Partial Seizures in Adult Tolerability Study (TS) Patients
Acronym: STARS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Was not possible to enroll sufficient number of subjects to draw any worthwhile conclusions from the study.
Sponsor: University of Pennsylvania (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 811542
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Complex Partial Seizures
Keywords: Tuberous sclerosis; TS; Seizures
MeSH Terms: conditions — Seizures; Tuberous Sclerosis | interventions — Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with Sabril (vigabatrin) (Other): This is a single arm study. All subjects who are eligible for treatment will begin taking vigabatrin (Sabril) during the third month of the study. Treatment will be in accordance with the FDA-approved prescribing information: upward titration will happen at a rate of 500mg per week until subjects reach their maximum tolerated dose, or 3g per day (whichever is lower). This dose may be decreased if needed under the supervision of the study doctor. Subjects who need to lower their dose or who stop taking Sabril will have their dosage decreased at a rate of 1 gm/week for one month under the supervision of the study doctor.
  Interventions: Drug: vigabatrin

INTERVENTIONS:
Drug: vigabatrin — Subjects will begin taking vigabatrin (Sabril) during the third month of the study. Upward titration will happen at a rate of 500mg per week until subjects reach their maximum tolerated dose, or 3g per day (whichever is lower). This dose may be decreased if needed under the supervision of the study doctor. Subjects who need to lower their dose or who stop taking Sabril will have their dosage decreased at a rate of 1 gm/week for one month under the supervision of the study doctor.
  Other Names: Sabril

SUMMARY:
This is an open-label, phase 4 study to examine the safety and efficacy of vigabatrin (Sabril) in Tuberous Sclerosis patients, a subset of the larger refractory complex partial epilepsy population for which the drug is approved. While enrolled on this trial, subjects will continue to take all of their normally prescribed medications, including their other antiepileptic drugs (AEDs).

Alternatively, there is a prospective observational arm that subjects who are about to take Sabril as treatment for seizures associated with Tuberous Sclerosis may join. Subjects who join this arm will not have any study visits and will not be asked to do anything specifically for the study. The study team will collect all study data from subjects' medical records only.

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's legally authorized representative must sign and date the Institutional Review Board approved Informed Consent and HIPPA Authorization Form.
* Male and female patients 18+ years of age with a clinical diagnosis of Tuberous Sclerosis who experience an average of at least three partial seizures every two months, of which one must be a complex partial seizure
* Patient must be on at least one and a maximum of four AEDs. Patient must be on a stable AED dose regimen for at least 30 days prior to screening. Neither a Vagal Nerve Stimulator (VNS) nor the ketogenic diet will count as an AED
* In the investigator's opinion, the patient or caregiver must be able to keep a seizure diary
* An MRI in the last 5 years, or willingness to undergo an MRI as part of the screening process

Exclusion Criteria:

* Cause of patient's seizures is a neurologic disease that is not Tuberous Sclerosis
* Current, clinical diagnosis of a major depressive episode or suicidal ideation
* Patient is taking more than four concurrent AEDs. Note: VNS or ketogenic diet is allowed and will not be counted in the four allowed AEDs
* Patient has a progressive CNS lesion confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan
* Patient is currently abusing drugs or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pollard, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for the treatment arm from within the Tuberous Sclerosis (TS) clinical at the University of Pennsylvania. Recruitment begain on 8/19/2010 and continued through 2013. All potential subjects had to be eligible to take Sabril (vigabatrin) under the FDA-approved prescribing information.
Pre-assignment Details: Before taking Sabril, subjects were required to undergo visual field and depression screenings in response to the FDA's black box warning about Sabril causing vision loss, and an increased risk of suicidal ideation among patients taking antiepileptic drugs like Sabril. No potential subjects were excluded due to screening assessments.
Groups:
- Treatment With Sabril (Vigabatrin): The interventional arm of this phase 4 study involved subjects taking vigabatrin (Sabril) in accordance with standard of care, FDA approved dosing instructions. There were no planned arms; all subjects followed the FDA-approved prescribing label.
  As there were not multiple treatment arms under investigation, per the FDA-approved prescribing label, the one and only subject who enrolled underwent upward titration happened at a rate of 500mg per week until she reached her maximum tolerated dose, or 3g per day. This dose was decreased as needed under the supervision of the study doctor. Again in accordance with standard of care, FDA-approved prescribing guidelines, when she stopped taking Sabril, her dosage decreased at a rate of 1 gm/week for one month under the supervision of the study doctor.
Period: Overall Study
Arm/Group | Treatment With Sabril (Vigabatrin)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Sabril (Vigabatrin): This is a single arm study. All subjects who are eligible for treatment will begin taking vigabatrin (Sabril) during the third month of the study. Treatment will be in accordance with the FDA-approved prescribing information: upward titration will happen at a rate of 500mg per week until subjects reach their maximum tolerated dose, or 3g per day (whichever is lower). This dose may be decreased if needed under the supervision of the study doctor. Subjects who need to lower their dose or who stop taking Sabril will have their dosage decreased by 1 gm/week for one month under the supervision of the study doctor.
Arm/Group | Treatment With Sabril (Vigabatrin)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [30 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Treatment: Female | 1
  Treatment: Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Safely Tolerating Sabril
Description: * Antiepileptic Drug (AED) levels in blood
  * Comprehensive panel (blood test)
  * Complete Blood Count with differential (blood test)
  * Visual field tests testing
  * Ophthalmology exam assessment
  * Frequency and severity of adverse events reported by subjects throughout their involvement with the study
Time Frame: Outcome measures will be assessed at the initiation of Sabril (titration), and at three and five months after starting Sabril. After this time, the subjects will have completed the study.
Population: One 30 year old female, Caucasian, non-Hispanic subject enrolled in the study. Due to adverse events, she did not complete the study, however, she completed all required follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Sabril (Vigabatrin)
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Patients Who Become Seizure Free While Taking Sabril
Description: * Seizure freedom
  * Responder rate (complex partial seizures only)
Time Frame: Seizure freedom will be assessed for the two month treatment phase of the study (months 4 and 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Sabril (Vigabatrin)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The study team used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | Treatment With Sabril (Vigabatrin)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Sabril (Vigabatrin) (N=1)
Seizure Cluster (Nervous system disorders) | 1 (2) — Subject was admitted to her local emergency room when she experienced seizure clusters that did not resolve with Diastat. SAE happened on twice.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Sabril (Vigabatrin) (N=1)
Fatigue (General disorders) | 1 (1)
seizures (Nervous system disorders) | 1 (1) — Increased seizure severity

LIMITATIONS AND CAVEATS:
The study was terminated due to insufficient enrollment; 98 potentially eligible patients were pre-screened and only one enrolled. The study was not terminated due to concerns regarding safety or efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No